CLINICAL TRIAL: NCT00644137
Title: Pregabalin Given to Tobacco Users to Study Addiction
Brief Title: GABA (Gamma Amino Butyric Acid) Medication for Tobacco
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0701002184; R01DA020752 (NIH); VA 0023 (Registry Identifier: VA); DPMC (Other: NIDA)
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Nicotine Dependence
Keywords: smoking sensations; no cravings; desire to smoke
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Pregabalin; Tobacco Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): pregabalin 300mg/day given in conjunction with smoking cigarettes.
  Interventions: Drug: pregabalin; Other: cigarettes
- 2 (Experimental): cigarettes given in conjunction with pregabalin
  Interventions: Drug: pregabalin; Other: cigarettes

INTERVENTIONS:
Drug: pregabalin — Help stop smoking
  Other Names: 300mg/day for pregabalin with smoking cigarettes
Other: cigarettes — help stop smoking with study medication

SUMMARY:
The goal of this study is to examine the effects of a GABA (gamma amino butyric acid)-enhancing medication, pregabalin (300 mg/day), on smoking behavior, tobacco withdrawal and cigarette craving in smokers. We hypothesize that in smokers, pregabalin at 300 mg/day, will be more effective than placebo in decreasing smoking behavior and attenuating tobacco withdrawal and cigarette craving.

DETAILED DESCRIPTION:
A total of 40 smokers will be randomly assigned to a sequence of treatment conditions: 300 mg/day pregabalin or placebo treatment. Each treatment condition will last 4 days, separated by 3 to 15 days of washout period. Smokers will have twice daily outpatient visits during the first 3 days and a test session on day 4. In each treatment period, smokers will abstain from smoking for 2.5 days, starting at 10 pm on Day 1 until the test session on Day 4. During the test sessions, measures of smoking behavior and tobacco withdrawal will be obtained.

Smoking is an important public health problem costing over 430,000 lives a year in this county alone. The first line-treatments, Nicotine Replacement Treatments (NRT) or bupropion, compared to placebo, approximately double the long-term success rate for smoking cessation. Given that there remains 46 million smokers in this country and over 70 percent of them interested in quitting smoking, development of new treatments for smoking cessation will have great public health implications.

Currently this protocol is complete with 24 completers. This study has been published. (April 2011)

ELIGIBILITY:
Inclusion Criteria:

* Female and male smokers, aged 18 to 55 years
* History of smoking daily for the past 12 months
* at least 15 cigarettes daily
* In good health as verified by medical history
* screening examination
* screening laboratory tests
* not pregnant as determined by pregnancy screening, nor breast feeding
* using acceptable birth control methods.

Exclusion Criteria:

* History of pregabalin allergy
* Use of psychotropic medication antidepressants, antipsychotics DSM-IV axis I diagnosis (schizophrenia, bipolar disorder, major depression
* Dependence or abuse of alcohol or any other illicit or prescription drugs
* current use of any other tobacco products, including smokeless tobacco
* history of seizures
* Inability to fulfill all scheduled visits and examination procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
We believe this medication will help people to stop smoking | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States